CLINICAL TRIAL: NCT04346680
Title: Intraoperative Adipose-Derived Stem Cells Administration During the Secondary Release (Neurolysis) of a Reconstructed Nerve
Brief Title: Intraoperative ADSC Administration During Nerve Release
Acronym: NEUROASC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mossakowski Medical Research Centre Polish Academy of Sciences (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Anna Sarnowska, Head of Translational Platform for Regenerative Medicine MRC, Mossakowski Medical Research Centre Polish Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/2015
Record Dates: First submitted 2019-10-15; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Neurotmesis of Peripheral Nerve (Disorder)
Keywords: ADSC; nerve release; neurolysis; stem cells; scar; peripheral nerves
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Procedure: ADSC administration

INTERVENTIONS:
Procedure: ADSC administration — The treated nerve will be identified and released. Scar tissue will be removed, and nerve fibers will be exposed. Prepared solutions of ADSC will be administered via microinjection with a 30-G needle along the released nerve fascicles, above and below the reconstructed area and around the adjacent tissue, which stayed in contact with the nerves.

SUMMARY:
The goal of the investigator's observational, nonrandomized, open label study is to investigate the safety and efficacy of autologous adipose derived mesenchymal cells (ADSC) transplantation into the individuals with faiure in reconstruction of peripheral nerves. ADSC will be used during a last-chance surgery (neurolysis, nerve release) on a previously reconstructed nerve. All enrolled patients will have a documented at least 2-years clinical and electrophisiological observation. Each patient will recive once 10 microinjections of ADSC along the injured nerve, directly after nerve neurolysis. Safety, adverse events and efficacy will be confirmed by clinical, elecrophisiological (EMG, Sensory Thyreshold) and DASH survey.

DETAILED DESCRIPTION:
The aim of the study will be an evaluation of undifferentiated Adipose-Derived Stromal/Stem Cells (ADSC) usage during a last-chance surgery (neurolysis, nerve release) on a previously reconstructed nerve. Patients who experienced failure of nerve reconstruction will be included in the study. During the revisional surgery, nerve fascicles will be released, and ADSCs will be isolated from harvested fat with enzymatic method in a standarized conditions. Cells will be administered through microinjections along the fascicles and around the adjacent tissues after external neurolysis. The follow-up will be continued at least 36 months.

ELIGIBILITY:
Inclusion Criteria:

* clinically definite failure nerve reconstructed patients
* lack of improvement after previous treatment
* without severe, unstable chronic diseases
* Polish citizens

Exclusion Criteria:

* INR > 2 before liposuction
* primary haematological disease, including hypercoagulable states
* previous/current history of neoplasm or comorbidity that could impact upon patient's survival
* pregnancy /lactation
* alcohol abuse, cocaine amphetamine, etc.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-04-23 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2022-06-23 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological improvement | 1 year
  Improvement in EMG - the appearance of activities in denervated muscles